CLINICAL TRIAL: NCT03478813
Title: Voiding School as a Treatment of Children's Functional Incontinence - Evaluation and Implementation of the Intervention
Brief Title: Voiding School as a Treatment of Children's Day-time Incontinence or Enuresis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was withdrawn because of too few eligible participants.
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Turku (Other); Southern Health and Social Care Trust (Other Government)
Responsible Party: Principal Investigator, Anneli Saarikoski, MNSc, RN, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Voiding School
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Daytime Wetting; Enuresis; Functional Incontinence
Keywords: Intervention; Implementation; Children; Urotherapy
MeSH Terms: conditions — Diurnal Enuresis; Enuresis

STUDY DESIGN:
Intervention Model Description: A parallel randomized trial conducted in 9 Child welfare clinics in one City in southern Finland. The study subjects are randomly allocated into intervention and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Voiding school (VS) is based on urotherapy guidelines for educating children with incontinence highlighting regular voiding habits and life-style advice. Learning by doing, understanding the body function by concrete example videos and pictures, and discussing are the main teaching methods.The intervention is delivered face-to-face in groups of 4-6 children. The VS includes three sessions one months apart. Duration of each VS session is three hours. The intervention is delivered with detailed manual. The intervention is provided by an urotherapist and a public-health nurse.
  Interventions: Behavioral: Voiding school
- Usual care group (No Intervention): The control group receives treatment according to the new 2016 guidelines of incontinence care in child welfare clinics in the city concerning. Treatment is carried out by public health nurse individually in consulting hours or by telephone.

INTERVENTIONS:
Behavioral: Voiding school — Children are educated on the kidneys, bladder and bowel function, the importance of regular voiding and drinking habits, and avoidance of constipation. Balloons, books, videos, animations, the pictures of a satisfied and irritated bladder and a poo-cars formula track are used to exemplify the function of urinary and defecation systems. During toilet visits children are given advise about an adequate and relaxed toilet posture with the help of little bench under the feet if needed. Each child also make their own timetable for peeing, pooing, and water drinking times, which they then should learn to follow in day-care, pre-school and at home. At the end of each session child, parent and public health nurse/urotherapist discuss any individual advice and the homework for the next time.
  Arms: Intervention group

SUMMARY:
The Voiding School is a simple educational intervention to treat children with daytime incontinence or enuresis.The purpose of this study is to implement the intervention in primary care, child welfare clinics. Half of the participated children will receive treatment according the Voiding School protocoll and half of them will receive treatment as usual. Patient outcomes are evaluated by measuring changes in wetting episodes. Aim is also to evaluate the implementation process.

DETAILED DESCRIPTION:
Children under school age attend to regular visits in Child welfare clinics for health examination and guidance. If the child have daytime incontinence or enuresis during the yearly visit at the age of 5 or 6, he or she is eligible for participating the study aiming to implement and evaluate the Voiding school intervention.

In the Voiding school the children are educated in groups of 4-6 children with child-oriented methods highlighting learning by doing in order to achieve better bladder control. Usual care includes individual advice concerning voiding habits and general life-style advice.

ELIGIBILITY:
Inclusion Criteria:

* The child is eligible for participating the study, if he or she has day-time incontinence or enuresis weekly, provided that following inclusion criteria are met: 1) there is no organic cause for incontinence, 2) he or she have no diagnosed behavioral disorders, and 3) the child and the parents are able to communicate in Finnish.

Exclusion Criteria:

* No specified exclusion criteria were set.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in wetting episodes | at baseline, after intervention (3 months), follow-up 6 months after baseline
  Changes of amount of dry days and nights, is performed with the modified Finnish version of the ICCS one-week voiding diary (©2015 International Children's Continence Society). Children with the help of their parents are asked to mark X in the diary every time they are voiding; M=a little amount of wetting, MM=a bigger amount of wetting, Y=night-time wetting. Bowel movements are marked with K.

SECONDARY OUTCOMES:
Changes in symptoms accosiated with incontinence | at baseline, after intervention (3 months), follow-up 6 months after baseline
  Symptom score for dysfunctional elimination syndrome (NLUT-DES questionnaire) is used to evaluate children's voiding and defecation habits associated with incontinence. It is a 14-item 5-point Likert scale questionnaire (0=no symptoms 4=severe symptoms, except item 3: 0=5-6 times, 2= 3-4 or 7-8 times, 4= 1-2 or over 8 times). Official translation into Finnish was performed for this study.
Changes in quality of life | at baseline, after intervention (3 months), follow-up 6 months after baseline
  Quality of life of 5-6 years old children with incontinence is measured with Finnish version of Pediatric Quality of Life Inventory (PedsQL™ 4.0) Used version is intended for parents of 5-7 years old children. Generic score scales (physical, emotional, social, school functioning) consist of 21-item 5-point Likert scale (0=never 4=always).

OTHER OUTCOMES:
Questionnaire of the background information of the child | at baseline
  Background information of the participated children (age, sex, dg, duration of incontinence, earlier treatment, constipation) is collected with developed questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Anneli Saarikoski, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Child welfare clinics, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
The data will be reported in articles including in summary of master thesis